CLINICAL TRIAL: NCT03741166
Title: Blood Collection Sub-Study of Exact Sciences Protocol 2018-10: "An Evaluation of a Multi-target Stool DNA (Mt-sDNA) Test, Cologuard, for CRC Screening in Individuals Aged 45-49 and at Average Risk for Development of Colorectal Cancer: Act Now"
Brief Title: Blood Collection Sub-Study for CRC Screening in Individuals 45-49 at Average Risk for CRC.
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-10B
Record Dates: First submitted 2018-10-31; First posted 2018-11-14 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Colo-rectal Cancer
Keywords: Blood Draw
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual blood samples may be used for evaluating performance of biomarkers for feasibility and assay development. Sample may be stored for up to 20 years. These blood samples will be de-identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject aged 45-49 with Average CRC Risk: Subjects will be men and women, 45-49 years of age, who enroll in Exact Sciences Protocol 2018-10. Subjects will provide a blood sample at time of enrollment.
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — Subjects participating in the study will have blood drawn at enrollment.

SUMMARY:
The primary objective of this sub-study, 2018-10B, is to collect blood specimens to assess new biomarkers for the detection of Colorectal Cancer (CRC).

DETAILED DESCRIPTION:
Subjects who consent to enroll in Exact Sciences Protocol 2018-10, will be asked to participate in this sub-study. Subjects enrolled in the Exact Sciences Protocol 2018-10, who provide written informed consent to participate in this sub-study, will have a blood sample collected at enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is currently enrolled in Exact Sciences Protocol 2018-10
2. Subject is willing and able to provide a blood sample.
3. Subject is willing and able to sign informed consent.

Exclusion Criteria:

1. Subject has any condition that in the opinion of the Investigator should preclude participation in the study.

Ages: 45 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be men and women, 45-49 years of age, who enroll in Exact Sciences Protocol 2018-10. Up to 942 subjects will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 871 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Blood-based biomarkers associated with genetic and epigenetic alterations. | Point in time blood collection (1 day) at enrollment
  Biomarkers under evaluation include differential methylation of nucleic acids and altered expression of proteins in blood from subjects at average risk for development of colorectal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Imperiale, Principal Investigator — Indiana University
Locations (37):
- United States (37):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Ventura County Gastroenterology, Camarillo, California
  - Alliance Research Centers, Laguna Hills, California
  - Focilmed, Oxnard, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Yale University Section of Digestive Diseases and Liver Diseases, New Haven, Connecticut
  - Precision Clinical Research, LLC, Lauderdale Lakes, Florida
  - Northshore University Health System Evanston Hospital, Evanston, Illinois
  - DM Clinical Research- Southwest Gastroenterology, Oak Lawn, Illinois
  - Deaconess Clinic- Mt. Pleasant, Evansville, Indiana
  - Deaconess Clinic- Gateway, Newburgh, Indiana
  - Johnson County ClinTrials, LLC, Lenexa, Kansas
  - New Orleans Research Institue, Metairie, Louisiana
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - Investigative Clinical Research, Annapolis, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - Capitol Research, Rockville, Maryland
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - United Medical Associates, Binghamton, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - Charlotte Gastroenterology & Hepatology, PLLC, Charlotte, North Carolina
  - Wilmington Gastroenterology Associates, Wilmington, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Comprehensive Internal Medicine, Inc., Wooster, Ohio
  - Family Practice Center of Wooster, Inc./Clinical Trial Developers, Wooster, Ohio
  - Gastroenterology Associates, PA, Greenville, South Carolina
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - University of Texas Health Science Center- McGovern Medical School, Houston, Texas
  - DM Clinical Research- PCP for Life, Houston, Texas
  - Virginia Gastroenterology Institute, Suffolk, Virginia
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after de-identification. This may include text, tables, figured, and appendices. The study protocol and informed consent form will also be shared. Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available from 2 years and ending 4 years after publication
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research.

DOCUMENTS (1):
  • Study Protocol (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT03741166/Prot_000.pdf